CLINICAL TRIAL: NCT01160887
Title: Is Diabetic Peripheral Neuropathy Accompanied by Internal Nerve Damage? A Comparative, Clinical Experimental Study of Peripheral and Visceral Nerve Damage in Diabetic Patients and Healthy Controls
Brief Title: Diabetes Peripheral Neuropathy and Small-fibre Nerve Damage: A Comparative Study
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/1652
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus; Peripheral Neuropathy; Small Fibre Neuropathy; Autonomic Neuropathy
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases; Small Fiber Neuropathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with diabetic peripheral neuropathy
- Healthy matched controls

SUMMARY:
The purpose of this study is to investigate whether patients with diabetes-related peripheral neuropathic pain also have non-recognized damage to the intestine caused by autonomic neuropathy. The model will shed light on aspects of peripheral nerve injuries on both somatic and as well as visceral sensory nerves. Classical autonomic parameters from electrocardiography (ECG) and Holter (24-h ECG and blood pressure) are compared with peripheral nerve injuries. The damage of autonomic nerves often recognized late in the course when patients develop gastroparesis, however an earlier recognition of this nerve damage may help clarifying the fundamental pathomechanisms and thereby optimize treatment for this patient group in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 18 and 75 years with diagnosed diabetes mellitus, according to WHO criteria (World Health Organization).
2. Proven peripheral neuropathy.
3. Oral and written consent, with documentation that all relevant information about the program is given to the patient.
4. The patient must be willing and able to, to meet the planned visit and meet the planned curriculum, including the participation in the experimental investigations.

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Medical or surgical disease for the study doctor's assessment makes the patient unsuitable for participation in the study
3. Previous or ongoing major depression
4. Patients who can or will not comply with the recommended instructions given by the study doctor
5. Use of analgesic opioid medication less than 24 hours before screening
6. Competitive conditions that can cause peripheral neuropathy (eg, herpes zooster)
7. Clinically significant disease less than 2 weeks from the planned entry in the study
8. People involved in the planning or execution of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with verified diabetic neuropathy.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
glucose | one year

CONTACTS AND LOCATIONS:
Overall Officials: Georg Dimcevski, MD, PhD, Principal Investigator — Haukeland University Hospital, Bergen, Norway
Locations (1):
- Haukeland University Hospital, Bergen, Norway